CLINICAL TRIAL: NCT03833700
Title: An Open-label Phase 1 Study of E7386 in Subjects With Advanced Solid Tumor Including Colorectal Cancer
Brief Title: A Study of E7386 in Participants With Advanced Solid Tumor Including Colorectal Cancer (CRC)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: E7386-J081-103
Record Dates: First submitted 2019-02-06; First posted 2019-02-07 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-01

CONDITIONS: Solid Neoplasms; Colorectal Neoplasms; Gastrointestinal Tumors
Keywords: Solid Tumor; Colorectal Cancer; E7386; Small Bowel Carcinoma; Gastrointestinal Neuroendocrine Tumor; Adrenocortical carcinoma; Desmoid Tumor; Solid pseudopapillary neoplasm of pancreas; Hepatocellular carcinoma
MeSH Terms: conditions — Colorectal Neoplasms; Digestive System Neoplasms; Gastro-enteropancreatic neuroendocrine tumor; Adrenocortical Carcinoma; Desmoid Tumors; Carcinoma, Hepatocellular | interventions — E-7386

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation Part: E7386 (Experimental): Participants will receive E7386 in 28-days treatment cycle until disease progression (PD), development of unacceptable toxicity, participant's request to discontinue, withdrawal of consent, or termination of the study program.
  Interventions: Drug: E7386
- Expansion Part 1 (Experimental): Participants will receive E7386 in 28-days treatment cycle until PD, development of unacceptable toxicity, participant's request to discontinue, withdrawal of consent, or termination of the study program.
  Interventions: Drug: E7386
- Expansion Part 2 (Experimental): Participants will receive E7386 in 28-days treatment cycle until PD, development of unacceptable toxicity, participant's request to discontinue, withdrawal of consent, or termination of the study program.
  Interventions: Drug: E7386

INTERVENTIONS:
Drug: E7386 — E7386 doses.

SUMMARY:
This study will be conducted to assess the safety and tolerability of E7386 in participants with solid tumor including CRC.

DETAILED DESCRIPTION:
The study will be conducted in 3 parts: dose escalation part, expansion part 1 and expansion part 2. The study will consist of Primary Assessment Phase and Continuation Phase. Primary Assessment Phase will include Pre-treatment Phase, Treatment Phase and Extension Phase (in expansion parts only).

After Treatment Phase, participants will be followed in follow-up period of Extension Phase (in expansion parts only). All participants who are still on study drug at the time of data cutoff date for the planned primary analysis will enter the Continuation phase and continue to receive E7386.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with a histological and/or cytological diagnosis of solid tumor must have any of the following tumor types:

   1. Dose Escalation Part: Participants with advanced, unresectable, or recurrent solid tumor including CRC for which no alternative standard therapy or no effective therapy exists
   2. Expansion Part 1: Participants with advanced, unresectable, or recurrent CRC in third- or later-line, Or participants with other gastrointestinal tumors such as small bowel carcinoma and gastrointestinal neuroendocrine tumors after at least 1 prior systemic chemotherapy regimen upon discussion and agreement with the sponsor
   3. Expansion Part 2: Participants with advanced, unresectable, or recurrent solid tumors expected to be highly dependent on wingless/integrated (Wnt)/β-catenin signaling pathway as specified below, who have no standard therapy. Disease progression must be confirmed within the past 12 months.

      * Desmoid tumor
      * Solid pseudopapillary neoplasm (SPN) of pancreas
      * Small bowel carcinoma with mutation of catenin beta-1 (CTNNB1) or adenomatous polyposis coli (APC)
      * Adrenocortical carcinoma (ACC) with mutation of CTNNB1, APC or zinc and ring finger 3 (ZNRF3)
      * Solid tumors (except for CRC) with APC mutation in participants diagnosed as familial adenomatous polyposis (FAP)
      * Hepatocellular carcinoma (HCC) with CTNNB1 gain-of-function mutation
      * Other types of solid tumors (except for CRC) harboring one or more Wnt-related gene mutations (example, APC, AXIN1, CTNNB1, ring finger protein 43 [RNF43], et cetera) expected to be highly dependent on Wnt/β-catenin signaling pathway based on emerging data may be enrolled upon consultation and agreement with the sponsor.

   HCC participants must have:
   1. A diagnosis of HCC that is histologically or cytologically confirmed (excluding fibrolamellar, sarcomatoid or mixed cholangio-HCC tumors) or clinically confirmed according to American Association for the Study of Liver Disease criteria, including cirrhosis of any etiology and/or chronic hepatitis B or C infection.
   2. Barcelona Clinic Liver Cancer (BCLC) Stage C disease, or BCLC Stage B disease not amenable to locoregional therapy or refractory to locoregional therapy, and not amenable to a curative treatment approach
2. Life expectancy of >=12 weeks.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
4. All AEs due to previous anti-cancer therapy have either returned to Grade 0-1 except for alopecia and Grade 2 peripheral neuropathy (renal/bone marrow/liver function should meet the inclusion criteria).
5. Adequate washout period before study drug administration:

   1. Chemotherapy and radiotherapy: 3 weeks or more
   2. Any therapy with antibody (Ab): 4 weeks or more
   3. Any investigational drug or device: 4 weeks or more
   4. Blood/platelet transfusion or Granulocyte-colony stimulating factor (G-CSF): 2 weeks or more
6. Adequate renal, bone marrow, liver function, and serum mineral level.
7. At least one measurable lesion based on RECIST 1.1.
8. Dose escalation part: Participants must consent to skin biopsies from skin tissue that is tumor-free during the study. Expansion part 1: At least 5 participants in each dose level must consent to skin biopsies from skin tissue that is tumor-free during the study. Participants may be enrolled without skin biopsies upon consultation and agreement by the sponsor. Expansion part 2: Participants must consent to skin biopsies from skin tissue that is tumor-free during the study in principle. Participants may be enrolled without consent to skin biopsies upon consultation and agreement by the sponsor.

Exclusion Criteria:

1. Known to be human immunodeficiency virus (HIV) positive.
2. Active infection requiring systemic treatment.

   For participants with HCC in Expansion part 2: In case of Hepatitis B surface antigen (HBsA g) positive (+) participants:
   1. Antiviral therapy for Hepatitis B virus (HBV) is not ongoing
   2. HBV viral load is 2000 International units per milliliter (IU/mL) or more at the Screening Period although antiviral therapy for HBV is ongoing
   3. Has dual active HBV infection (HBsAg [+] and/or detectable HBV Deoxyribonucleic acid [DNA]) and Hepatitis C virus (HCV) infection (anti-HCV Ab [+] and detectable HCV Ribonucleic acid [RNA]) at study entry
3. Diagnosed with meningeal carcinomatosis.
4. Participants with brain or subdural metastases are not eligible, unless they have completed local therapy and have discontinued the use of corticosteroids for this indication for at least 4 weeks before starting treatment in this study. Any signs (example: radiologic) or symptoms of brain metastases must be stable for at least 4 weeks before starting study treatment.
5. Pulmonary lymphangitic involvement that results in pulmonary dysfunction requiring active treatment, including the use of oxygen.
6. Any of bone disease/conditions as follows;

   1. Osteoporosis with T-score less than (<) -3 at the left or right total hip, left or right femoral neck or lumbar spine (L1-L4) as determined by dual energy X-ray absorptiometry (DXA) scan. Participants with T-score <-2.5 to -3.0 and no prior medical therapy for osteoporosis can only be included provided that treatment with a bisphosphonate (example, zoledronic acid) or denosumab has been started at least 14 days prior to the first dose of study drug
   2. Metabolic bone disease, such as hyperparathyroidism, Paget's disease or osteomalacia
   3. Symptomatic hypercalcemia requiring bisphosphonate therapy
   4. History of any fracture within 6 months prior to starting study drug
   5. Any condition requiring orthopedic intervention
   6. Bone metastasis, not being treated by bisphosphonate or denosumab. Participant may be included if treatment with bisphosphonate or denosumab have been started at least 14 days prior to the first dose of study drug. Participants with previous solitary bone lesions controlled with radiotherapy are eligible
   7. History of symptomatic vertebral fragility fracture or any fragility fracture of the hip, pelvis, wrist or other location (defined as any fracture without a history of trauma or because of a fall from standing height or less)
   8. Moderate (25 percent [%] to 40% decrease in the height of any vertebrae) or severe (more than [>] 40% decrease in the height of any vertebrae) morphometric vertebral fracture at baseline.
7. History of active malignancy (except for original disease, or definitively treated melanoma in-situ, basal or squamous cell carcinoma of the skin, carcinoma in-situ of the bladder or cervix, or early stage gastric/colorectal cancer) within the past 24 months prior to the first dose of study drug.
8. For participants with HCC in Expansion part 2, if the participants have:

   1. Child-Pugh status of B and C
   2. History of hepatic encephalopathy within 6 months prior to starting study drug unresponsive to therapy within 3 days. Participants on rifaximin or lactulose during screening to control their hepatic encephalopathy are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-03-05 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose-limiting Toxicities (DLTs) | Baseline up to Cycle 1 (Cycle length is equal to [=] 28 days)
  DLT will be defined as any of the events that are considered by the investigator to be at least possibly related to therapy with the study medication. Toxicity will be evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE 5.0).
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 30 days after the last dose of study drug or before initiating post anti-cancer treatment (approximately 6 years)

SECONDARY OUTCOMES:
Cmax: Maximum Observed Plasma Concentration for E7386 | Dose escalation Part, Cycles 1 to 6: Up to Day 8; Dose Expansion Part 1 and 2, Cycles 1 and 2: Up to Day 8 (Cycle length=28 days)
Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for E7386 | Dose escalation Part, Cycles 1 to 6: Up to Day 8; Dose Expansion Part 1 and 2, Cycles 1 and 2: Up to Day 8 (Cycle length=28 days)
AUC: Area Under the Plasma Concentration Versus Time Curve for E7386 | Dose escalation Part, Cycles 1 to 6: Up to Day 8; Dose Expansion Part 1 and 2, Cycles 1 and 2: Up to Day 8 (Cycle length=28 days)
CL/F: Apparent Total Body Clearance for E7386 | Dose escalation Part, Cycles 1 to 6: Up to Day 8; Dose Expansion Part 1 and 2, Cycles 1 and 2: Up to Day 8 (Cycle length=28 days)
Vz/F: Apparent Volume of Distribution for E7386 | Dose escalation Part, Cycles 1 to 6: Up to Day 8; Dose Expansion Part 1 and 2, Cycles 1 and 2: Up to Day 8 (Cycle length=28 days)
Objective Response Rate (ORR) | From first dose of study drug until PD, development of unacceptable toxicity, participant requests to discontinue, withdrawal of consent or study termination (up to approximately 6 years)
  The ORR is defined as the percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR). The ORR will be assessed by investigator based on RECIST version 1.1.
Disease Control Rate (DCR) | From first dose of study drug until PD, development of unacceptable toxicity, participant requests to discontinue, withdrawal of consent or study termination (up to approximately 6 years)
  DCR is defined as the percentage of participants with a BOR of CR, PR, or stable disease (SD). The DCR will be assessed by investigator based on RECIST version 1.1.
Clinical Benefit Rate (CBR) | From first dose of study drug until PD, development of unacceptable toxicity, participant requests to discontinue, withdrawal of consent or study termination (up to approximately 6 years)
  The CBR is defined as the percentage of participants with a BOR of CR, PR, or durable SD. The CBR will be assessed by investigator based on RECIST version 1.1.
Progression-free Survival (PFS) | From first dose of study drug until PD, or death from any cause, whichever occurs first (up to approximately 6 years)
  PFS is defined as the time from the date of the first dose to the date of the first documentation of confirmed PD or death, whichever occurs first.
Duration of Response (DOR) | From the date of first documented CR or PR until first documentation of PD or death (up to approximately 6 years)
  DOR is defined as the time from the first date of documented CR or PR to the date of PD or death, whichever occurs first. It will be calculated for participants whose BOR is CR or PR. DOR will be assessed according to RECIST version 1.1.
Overall Survival (OS) | From first dose of study drug until date of death (up to approximately 6 years)
  OS is defined as the time from the date of first dose to the date of death.

CONTACTS AND LOCATIONS:
Locations (8):
- Japan (8):
  - Eisai Trial Site#7, Nagoya, Aichi-ken
  - Eisai Trial Site #2, Kashiwa, Chiba
  - Eisai Trial Site #5, Sapporo, Hokkaido
  - Eisai Trial Site#8, Sendai, Miyagi
  - Eisai Trial Site #3, Nagaizumi-cho, Shizuoka
  - Eisai Trial Site #1, Chuo Ku, Tokyo
  - Eisai Trial Site #4, Fukuoka
  - Eisai Trial Site#6, Osaka

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.